CLINICAL TRIAL: NCT05656287
Title: My Mobile Wallet: An Intervention to Support Access to Tuberculosis Care and Medication Adherence in Rural Uganda
Brief Title: My Mobile Wallet: An Intervention for Tuberculosis Medication Adherence in Rural Uganda
Acronym: M_wallet
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUST-2021-102
Record Dates: First submitted 2022-09-20; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; mobile health; mobile money; adherence
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: Participants will be randomized using the 1:1:1 allocation ratio to the following arms: 1) SMS + incentives (Arm A) 2) SMS only (Arm B), and 3) no SMS (control). All participants will have adherence monitored in real-time for 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): (Arm A): For the first two months, 54 participants will receive i) daily SMS medication reminders, ii) monthly mobile money for transport to the clinic, and iii) monthly mobile money incentives if >90% medication adherence. For the remaining four months, the participants will receive: i) weekly medication SMS reminders, ii) monthly mobile money for transport to the clinic, iv) monthly mobile money incentives if >90% medication adherence.
  Interventions: Other: SMS texts + incentives + Wisepill device for medication monitoring
- Arm B (Experimental): For the first 2 months, 54 participants will receive daily SMS medication reminders, ii). For the remaining 4 months, the participants will receive weekly medication SMS reminders.
  Interventions: Other: SMS texts only + Wisepill device for medication monitoring
- Arm C- Control (Experimental): Participants (54) in the Control (Arm C) will not receive SMS reminders or mobile money
  Interventions: Other: Wisepill device for medication monitoring only

INTERVENTIONS:
Other: SMS texts + incentives + Wisepill device for medication monitoring — For the first two months, 54 participants will receive i) daily SMS medication reminders, ii) monthly mobile money for transport to the clinic, and iii) monthly mobile money incentives if >90% medication adherence. For the remaining four months, the participants will receive: i) weekly medication SMS reminders, ii) monthly mobile money for transport to the clinic, iv) monthly mobile money incentives if >90% medication adherence.
  Arms: Arm A
Other: SMS texts only + Wisepill device for medication monitoring — For the first 2 months, 54 participants will receive daily SMS medication reminders, ii). For the remaining 4 months, the participants will receive weekly medication SMS reminders. All participants will also receive a Wisepill device for medication monitoring.
  Arms: Arm B
Other: Wisepill device for medication monitoring only — Participants (54) in the Control arm will not receive SMS reminders or mobile money. All participants will also receive a Wisepill device for medication monitoring.
  Arms: Arm C- Control

SUMMARY:
The goal of this clinical trial is to develop My Mobile Wallet- a behavioral and economic intervention to support tuberculosis treatment adherence in rural southwestern Uganda. The main question[s] it aims to answer are: • Determine the optimal design and develop My Mobile Wallet as an intervention to support tuberculosis medication adherence • Assess the initial feasibility and acceptability of using My Mobile Wallet to support tuberculosis medication. Participants will use My Mobile Wallet intervention for a period of six months. Researchers will compare My Mobile Wallet intervention versus standard care to see if there is an impact on tuberculosis medication adherence.

DETAILED DESCRIPTION:
Tuberculosis is a serious public health concern which kills more people annually than HIV and malaria combined. Worldwide, nearly 10 million people develop tuberculosis and nearly 2 million people die from tuberculosis annually. Low-income countries account for more than 90% of tuberculosis cases and deaths. Uganda faces a high burden of tuberculosis with a prevalence rate of 253 per 100,000 people and an incidence rate of 201 per 100,000 people. Additionally, tuberculosis is a leading cause of death among individuals living with HIV/AIDS.

Poor treatment adherence limits the success of tuberculosis treatment and increases tuberculosis transmission. The treatment success rate in Uganda stands at 75%, below the national target of 90%. Poor tuberculosis medication adherence can lead to treatment failure, development of drug-resistant TB, and secondary transmission. Importantly, treatment for multi-drug resistant (MDR) tuberculosis is difficult to tolerate, prolonged, and expensive.

Uganda currently spends US$105 (on transport refund and food incentives) per month on each MDR-TB patient from the time they are discharged (after the initial six months of hospitalization) until treatment completion (one year). This translates to a cost of $1,260 per patient for the 12 months of treatment. Currently, Uganda has about 16,000 MDR-TB patients. The My Mobile Wallet intervention supports treatment adherence, potentially preventing drug resistance, thereby relieving the country of the financial burden associated with MDR-TB treatment. Importantly, treatment for MDR-TB is difficult to tolerate, prolonged, and leads to productivity loss for patients and their caregivers, which negatively affects the economic development of the country.

Socio-economic determinants of health are a major driver of tuberculosis infection and non-adherence. Although tuberculosis treatment that works well has existed since the 1940s, many people delay seeking treatment, struggle with medication adherence, and/or do not complete their treatment because of behavioral and socio-economic factors. Preliminary data from the ongoing K43 (K43TW010388) study indicate that financial insecurity constrains medication adherence. Tuberculosis leads to the loss of productivity of patients and their caregivers, resulting in additional costs for patients (e.g., in form of transport to the clinic), and may lead to loss of employment for fear of spreading the disease to other people.

Moreover, having tuberculosis is associated with other negative socioeconomic consequences, such as divorce, school interruptions for children, and social exclusion, in addition to the hardship of deteriorating health. Currently in Uganda, 53% of tuberculosis patients take loans and/or sell property to meet the costs of their tuberculosis care. Two in every 10 people (21% of the population) live on $1.25 a day or less in Uganda, making saving for health difficult amidst other immediate competing interests. Because tuberculosis disproportionately affects the poorest in the population, its poverty-aggravating effects are felt more by those who are already vulnerable. Interventions are necessary to overcome the poverty-based structural barriers to tuberculosis treatment, including unconditional transportation to clinic.

Despite the great potential of financial incentives in improving tuberculosis care, research to date is limited, remains largely inconclusive, and has mainly focused on high- and middle-income countries, where financial incentives may have less effect. The World Health Organization End Tuberculosis strategy recommends using reimbursements and social protection schemes to lower the social and economic burden of tuberculosis and address social determinants of health. Although literature in this area is limited, a monthly financial incentive package improved tuberculosis treatment success and reduced loss to follow-up among poor people in Nigeria.

A literature review indicates that cash transfer interventions for patients in low- and middle-income countries initiating tuberculosis treatment may improve clinical outcomes. This review notes that to date, there is limited research utilizing incentives in tuberculosis care, findings from the modest existing research remain largely inconclusive, and research has mainly focused on high- and middle-income countries, where tuberculosis is not a priority, and where financial incentives may have less effect. For instance, in Brazil, cash transfers improved rates of tuberculosis cure by 82.1%. However, these studies use face-to-face approaches to provide incentives, which may be limited by geographical boundaries, are time consuming, and involve transport costs. My Mobile Wallet will provide opportunities for patients in low resource settings to electronically receive and spend money for TB-related treatment.

Rapidly expanding cellular networks across sub-Saharan Africa have greatly increased the capacity of cellular technology to serve as a novel solution to challenges and barriers in the tuberculosis epidemic. Cellular networks are becoming ubiquitous globally. According to Global System for Mobile Communications real-time intelligence data, there are currently over 5.1 billion people with mobile devices, and 8.97 billion mobile connections which exceeds the current world population of 7.7 billion. In Uganda specifically, mobile phone reception is available across the vast majority of the country, including many rural areas and among economically disadvantaged populations. A recent study from Uganda indicates that most tuberculosis patients (75%) own mobile phones and are willing to received TB-related support using mobile phones.

The use of mobile money-based approaches in low resource settings has shown considerable utility in the business sector and holds promise for health. The rapid evolution of mobile phones has enabled a mobile payment platform (often known as mobile money) which enables micro-banking financial transactions (e.g. sending, saving, paying, and receiving money) possible using simple mobile phones that are independent of Smartphone capabilities or internet access. Many people in Uganda are increasingly relying on mobile money as they lack access to formal banking services-more than 23.5 million people have mobile money subscriptions. The use of mobile money in rural areas has enabled farmers to address market failures, access financial services, pay utility bills, and settle supply costs, thus, unlocking opportunities to reach the underserved populations.

The use of mobile money for saving and making payment for pregnancy-related care was beneficial and feasible among pregnant women in Madagascar. Among hard-to-reach populations, mobile money has helped enable routine payment of health insurance and improve access to family planning. However, there is lack of evidence around mobile money to support tuberculosis treatment adherence.

Tuberculosis medication adherence interventions that work well in low resource settings to date are limited; however, SMS-based interventions show promise. The directly observed therapy (DOT) strategy recommended by the World Health Organization, which requires that patients take their medication under physical supervision, has been abandoned by many clinics in Uganda, as it demands a significant time commitment from health workers and treatment supporters, generates substantial financial burdens, and inhibits patient autonomy. The World Health Organization End Tuberculosis Strategy 2017 suggests a suite of new interventions to improve adherence, including mobile phone-based short message service (SMS) messages.

The use of SMS in addressing tuberculosis medication adherence challenges in low-resource settings to date are limited. The prevailing SMS-based studies for tuberculosis medication adherence report mixed results, and have largely been implemented in developed countries, leaving little known about limited-resource countries, heavily burdened by TB. The formative findings from an on-going K43 (K43TW010388) show that SMS may provide acceptable alternative approaches to supporting tuberculosis medication. The effects of these SMS reminders could be greater if combined with economic incentives. No study has assessed the use of SMS linked with economic incentives in supporting tuberculosis medication adherence.

Adherence interventions based on real-time electronic monitoring are feasible, acceptable, have shown to improve HIV treatment adherence. The investigators demonstrated the feasibility, acceptability, and impact on adherence of cellular technology for HIV medication adherence in rural Uganda. The current real-time tuberculosis adherence monitoring intervention the investigators are assessing (K43TW010388) has promise for addressing additional barriers in social support and habit formation. For example, findings indicate that real-time adherence monitoring technology serves as a reminder for both tuberculosis and HIV treatment among co-infected patients. However, financial barriers remain. Thus, combining SMS, mobile money incentives, and real-time monitoring has the potential to overcome the majority of tuberculosis adherence barriers.

Client-centered design increases the likelihood of the intervention uptake and use, as the end user is centrally involved in the development process. Failure to target approaches to local needs and norms limit the utility of health technologies in low-resource settings. Most strategies involve a user interface, therefore, reversing this trend will require behavioural and social science evaluation of acceptability and use of novel technologies in target populations.

Summary: Tuberculosis is a serious public health concern which kills more people annually than HIV and malaria combined. Poor treatment adherence limits the success of tuberculosis treatment and increases tuberculosis transmission. SMS and real-time adherence monitoring may provide low-cost and acceptable alternative approaches to supporting tuberculosis medication especially in settings where DOT is difficult to implement. Financial incentives have shown promise for improving tuberculosis care, but the approach has mainly been implemented in countries where tuberculosis is not a public health priority; moreover, current approaches require costly face-to-face interaction. My Mobile Wallet is a novel intervention that use SMS to remind patients to take their medication, as well as sending mobile money to cover transport costs to tuberculosis clinic, and motivate medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with TB per the clinic records (TB patients living with HIV will also be eligible)
* Starting TB treatment now or been on TB treatment for <2 weeks
* Owning a mobile phone
* Aged 18 years and older
* Live in Mbarara District
* Willing to grow hair on the head and to allow a small thatch of it/hair (10-25 strands/0.02 ng/mg) to be cut at month 2 and 4 in the study
* Willing and able to give consent.

Exclusion Criteria:

* Unable to use mobile money-based SMS (train and test this skill at recruitment)
* Severe mental condition limiting the ability to provide consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Medication adherence rates among patients | 6 months
  Number of patients in the intervention arm with higher adherence as electronically ascertained by the Wisepill device

SECONDARY OUTCOMES:
Number of patients who used the intervention | 6 months
  % of participants who used the intervention and reported technical problems. The intervention will be considered feasible if >70% participants 1) receive mobile money, 2) utilize the transport incentive for transport to the clinic, 3) receive SMS reminders
TB treatment completion | 6 months
  Number of patients who complete TB medication as ascertained by Medical records at the end of six months.
Clinic Attendance | 6 months
  Number of patients with continuous hospital attendance by reviewing the TB clinic medical records and My Mobile wallet intervention.
Mortality | 6 months
  Mortality rate as ascertained by medical records at the end of six months.
Cure rate | 6 months
  Number of patients cured as ascertained by medical records from the TB clinic at the end of six months

CONTACTS AND LOCATIONS:
Overall Officials: Angella Musiimenta, PhD, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara Regional Referral Hospital, Mbarara, Uganda

REFERENCES:
- [Background] World Health Organisation., Global tuberculosis control: WHO report 2000, in Global tuberculosis control:WHO report 2000. 2000.
- [Background] Horsburgh CR Jr, Barry CE 3rd, Lange C. Treatment of Tuberculosis. N Engl J Med. 2015 Nov 26;373(22):2149-60. doi: 10.1056/NEJMra1413919. No abstract available. PMID 26605929
- [Background] Adane AA, Alene KA, Koye DN, Zeleke BM. Non-adherence to anti-tuberculosis treatment and determinant factors among patients with tuberculosis in northwest Ethiopia. PLoS One. 2013 Nov 11;8(11):e78791. doi: 10.1371/journal.pone.0078791. eCollection 2013. PMID 24244364
- [Background] MOH, Direct and Indirect costs due to Tuberculosis and proportion of Tuberculosis-affected households experiencing catastrophic costs due to TB in Uganda. Ministry of Health Uganda. 2019.
- [Background] Musiimenta A, Tumuhimbise W, Mugaba AT, Muzoora C, Armstrong-Hough M, Bangsberg D, Davis JL, Haberer JE. Digital monitoring technologies could enhance tuberculosis medication adherence in Uganda: Mixed methods study. J Clin Tuberc Other Mycobact Dis. 2019 Aug 29;17:100119. doi: 10.1016/j.jctube.2019.100119. eCollection 2019 Dec. PMID 31788561
- [Background] Heil SH, Higgins ST, Bernstein IM, Solomon LJ, Rogers RE, Thomas CS, Badger GJ, Lynch ME. Effects of voucher-based incentives on abstinence from cigarette smoking and fetal growth among pregnant women. Addiction. 2008 Jun;103(6):1009-18. doi: 10.1111/j.1360-0443.2008.02237.x. PMID 18482424
- [Background] Charness, G. and U. Gneezy, Incentives to exercise. Econometrica, 2009. 77(3): p. 909-931.
- [Background] Linnemayr S, Stecher C. Behavioral Economics Matters for HIV Research: The Impact of Behavioral Biases on Adherence to Antiretrovirals (ARVs). AIDS Behav. 2015 Nov;19(11):2069-75. doi: 10.1007/s10461-015-1076-0. PMID 25987190
- [Background] Richterman A, Steer-Massaro J, Jarolimova J, Luong Nguyen LB, Werdenberg J, Ivers LC. Cash interventions to improve clinical outcomes for pulmonary tuberculosis: systematic review and meta-analysis. Bull World Health Organ. 2018 Jul 1;96(7):471-483. doi: 10.2471/BLT.18.208959. Epub 2018 Jun 4. PMID 29962550
- [Background] Torrens AW, Rasella D, Boccia D, Maciel EL, Nery JS, Olson ZD, Barreira DC, Sanchez MN. Effectiveness of a conditional cash transfer programme on TB cure rate: a retrospective cohort study in Brazil. Trans R Soc Trop Med Hyg. 2016 Mar;110(3):199-206. doi: 10.1093/trstmh/trw011. PMID 26884501
- [Background] Ggita JM, Ojok C, Meyer AJ, Farr K, Shete PB, Ochom E, Turimumahoro P, Babirye D, Mark D, Dowdy D, Ackerman S, Armstrong-Hough M, Nalugwa T, Ayakaka I, Moore D, Haberer JE, Cattamanchi A, Katamba A, Davis JL. Patterns of usage and preferences of users for tuberculosis-related text messages and voice calls in Uganda. Int J Tuberc Lung Dis. 2018 May 1;22(5):530-536. doi: 10.5588/ijtld.17.0521. PMID 29663958
- [Background] Ware NC, Idoko J, Kaaya S, Biraro IA, Wyatt MA, Agbaji O, Chalamilla G, Bangsberg DR. Explaining adherence success in sub-Saharan Africa: an ethnographic study. PLoS Med. 2009 Jan 27;6(1):e11. doi: 10.1371/journal.pmed.1000011. PMID 19175285
- [Background] Haberer JE, Musiimenta A, Atukunda EC, Musinguzi N, Wyatt MA, Ware NC, Bangsberg DR. Short message service (SMS) reminders and real-time adherence monitoring improve antiretroviral therapy adherence in rural Uganda. AIDS. 2016 May 15;30(8):1295-300. doi: 10.1097/QAD.0000000000001021. PMID 26760452
- [Background] Atukunda EC, Musiimenta A, Musinguzi N, Wyatt MA, Ashaba J, Ware NC, Haberer JE. Understanding Patterns of Social Support and Their Relationship to an ART Adherence Intervention Among Adults in Rural Southwestern Uganda. AIDS Behav. 2017 Feb;21(2):428-440. doi: 10.1007/s10461-016-1559-7. PMID 27671479
- [Background] Campbell JI, Aturinda I, Mwesigwa E, Burns B, Santorino D, Haberer JE, Bangsberg DR, Holden RJ, Ware NC, Siedner MJ. The Technology Acceptance Model for Resource-Limited Settings (TAM-RLS): A Novel Framework for Mobile Health Interventions Targeted to Low-Literacy End-Users in Resource-Limited Settings. AIDS Behav. 2017 Nov;21(11):3129-3140. doi: 10.1007/s10461-017-1765-y. PMID 28421356
- [Background] Linnemayr, S., Consumption smoothing and HIV/AIDS: The case of two communities in South Africa. Economic Development and Cultural Change, 2010. 58(3): p. 475-506.
- [Background] Linnemayr S, Glick P, Kityo C, Mugyeni P, Wagner G. Prospective cohort study of the impact of antiretroviral therapy on employment outcomes among HIV clients in Uganda. AIDS Patient Care STDS. 2013 Dec;27(12):707-14. doi: 10.1089/apc.2013.0139. PMID 24320014
- [Background] Linnemayr S, Lawson BS, Glick P, Wagner G. Economic Status and Coping Mechanisms of Individuals Seeking HIV Care in Uganda. J Afr Econ. 2011 Jun;20(3):505-529. doi: 10.1093/jae/ejr014. Epub 2011 May 4. PMID 35722172
- [Derived] Musiimenta A, Tumuhimbise W, Atukunda E, Mugaba A, Linnemayr S, Haberer J. Digital Adherence Technologies Linked to Mobile Money Incentives for Medication Adherence Among People Living With Tuberculosis: Mixed Methods Feasibility and Acceptability Study. JMIR Hum Factors. 2024 May 31;11:e47996. doi: 10.2196/47996. PMID 38819905
- [Derived] Musiimenta A, Tumuhimbise W, Atukunda E, Mugaba A, Linnemayr S, Haberer J. Digital Adherence Technologies and Mobile Money Incentives for Management of Tuberculosis Medication Among People Living With Tuberculosis: Mixed Methods Formative Study. JMIR Form Res. 2023 Apr 12;7:e45301. doi: 10.2196/45301. PMID 37043263